CLINICAL TRIAL: NCT04681534
Title: A Double-blind Crossover Study to Evaluate the Safety and Efficacy of Adaptive Deep Brain Stimulation Delivered Through AlphaDBS System in Patients With Parkinson's Disease
Brief Title: Safety and Efficacy of Adaptive Deep Brain Stimulation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Newronika (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NWK_AlphaDBS_FIM_2019
Record Dates: First submitted 2020-11-20; First posted 2020-12-23 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- conventional DBS (Active Comparator)
  Interventions: Device: AlphaDBS System
- adaptive DBS (Experimental)
  Interventions: Device: AlphaDBS System

INTERVENTIONS:
Device: AlphaDBS System — AlphaDBS can be programmed with two different types of stimulation: conventional DBS and adaptive DBS, that automatically adjusts the energy delivered to patient using a biosignal, local field potential (LFP), in a close loop configuration.

SUMMARY:
The aim of this study is to assess the safety and the potential efficacy of personalized Local Field Potential (LFP)-based adaptive Deep Brain Stimulation (aDBS), using the implantable pulse generator (IPG) of the "AlphaDBS" System, in Parkinson's Disease patients, chronically implanted in subthalamic nucleus (STN) for DBS.

DETAILED DESCRIPTION:
The study protocol is organized in two phases: the "short-term follow-up" and the "long-term follow-up".

PD patients in need of IPG replacement or "de novo DBS" patients will be screened for enrollment eligibility.

For the "short-term follow-up", randomized patients will undergo 2 days of experimental sessions (i.e. one per each type of stimulation mode, cDBS and aDBS), in a well-controlled environment (i.e. during hospitalization). This part of the study will collect information on safety and potential efficacy endpoints as assessed by experienced neurologists. The "short term follow-up" phase will be considered complete when the endpoint assessment has been performed for all patients.

Patients, who will not experience severe side effects and who will be deemed suitable by the neurologist, will be eligible to continue in the "long-term follow-up" phase (i.e. 1 month) in their "home" environment. The "AlphaDBS" System will deliver the stimulation in aDBS or cDBS mode, for two weeks in each mode.

ELIGIBILITY:
IPG Replacement Patients:

Inclusion Criteria

1. Diagnosis of idiopathic PD;
2. Subject is bilaterally treated with DBS in the STN using a Medtronic Activa PC or Activa RC IPG (mono-channnel or dual channel);
3. DBS implant for at least 3 years and in need of battery replacement within 12 months after consent;
4. Patients must be able to understand and sign the informed consent document.

Exclusion criteria

1. Patients with severe cognitive decline, as resulting from MoCA assessment (MoCA score < 10);
2. Patients with major psychiatric issues or any other condition that, based on the physician opinion, could interfere with the study conduct (e.g. severe depression, psychosis, etc.);
3. Patients with any medical conditions potentially interfering with DBS battery replacement surgery (e.g. severe hypertension, active cancer, intake of drugs interfering with the coagulation etc.);
4. Need to replace or reposition the leads during the IPG replacement procedure;
5. Patients with > 10 recurrent falls experienced in the 3 months prior to consent;
6. Patients that cannot tolerate an interruption of DBS stimulation for at least 30 min;
7. Patients taking less than one levodopa dose per day;
8. Patients without suitable LFPs recordings or with significant artifacts;
9. Pregnant or breastfeeding women.

De Novo DBS Patients:

Inclusion Criteria

1. Patient is ≥ 18 years old;
2. Patient has been diagnosed with levodopa-responsive idiopathic Parkinson's disease for ≥ 5 years;
3. The disease stage is II, III or IV according to the Hoehn and Yahr scale
4. Patient has history of improvement of PD-related symptoms as a direct result of levodopa intake;
5. Patient has been selected for bilateral STN or GPi DBS, independently from this study, in accordance with local standard of care DBS screening;
6. Patient has been selected to receive Medtronic leads model 3389 or 37086 or Abbott directional leads model number 6170 or 6172 or 6371, independently from this study, in accordance with local standard of care for DBS;
7. Patient has DBS-leads circuit integrity assessed and confirmed by impedance testing, before IPG implantation;
8. MoCA score > 26 in best medical condition;
9. BDI-II score < 17 in best medical condition;
10. UPDRS-III improvement by ≥ 33% with levodopa challenge test (at approximately 90 min from the intake of the usual morning levodopa dose plus 30%);
11. Patient is able to understand the study requirements and the treatment procedures and has provided written informed consent to participate;
12. Patient has a responsible caregiver who will help completing the 3-day diary, provide feedback on activities of daily living (ADL), and ensure the patient complies with visit schedule;
13. Patient is on stable PD-medication for one month prior surgery;
14. Patient is willing and able to attend all study-required visits, complete the study procedures and attend appropriate follow up visits.

Exclusion Criteria

1. Patient has contraindications for DBS surgery, including any intracranial abnormality (e.g., generalized atrophy, vascular malformation, hydrocephalus, hematoma, cavernous or venous angioma, tumor or metastases, midline shift, etc.) or metallic implant (e.g., aneurysm clip, cochlear implant, etc.);
2. Patient has a history of suicide attempt or current active suicidal ideation as determined by a positive response to Item 2-5 of suicide ideation sub-scale of the Columbia Suicide Severity Rating Scale (C-SSRS);
3. Patient has dementia, major depression, seizures, congestive heart failure, uncontrolled diabetes, dialysis, substance use disorders as described in DSM-V, or any other severe medical condition;
4. Patient has any medical condition that could interfere with study procedures, confound the assessment of study endpoints, or prevent a proper data collection;
5. Patient had confirmation of diagnosis of a terminal illness associated with survival < 12 months;
6. Patient needs repeated MRI scans;
7. Patient requires diathermy, transcranial magnetic stimulation (TMS), or electroconvulsive therapy (ECT);
8. Patient carries an electrical or electromagnetic implant (e.g., cochlear prosthesis, pacemaker, neurostimulator, etc.);
9. Patient has, or plans to obtain, an implanted electrical stimulation medical device and/or an implanted medication pump (e.g., DUOPATM infusion pump) and/or is treated with a portable infusion pump;
10. Patient is on anticoagulant therapy which cannot be paused for > 5 days before IPG implant surgery;
11. Patient with a history of cranial surgery including ablation procedure or any other previous neurosurgical procedure for the treatment of PD symptoms on either side of the brain;
12. Patient is currently participating in another clinical study (excluding any sub-study of the present study);
13. Patient is a female who is breastfeeding or of child-bearing potential with a positive urine pregnancy test or not using adequate contraception;
14. Patients without suitable LFPs recordings or with significant artifacts.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-01-26 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of the "AlphaDBS" System, when used in cDBS and aDBS mode | 1 month
  Occurrence of device related adverse events

SECONDARY OUTCOMES:
PD-related motor symptoms and their fluctuations | 1 month
  Evaluation of PD-related motor symptoms using the Unified Parkinson's Disease Rating Scale - UPDRS Part III.
Dyskinesia | 1 month
  Evaluation of dyskinesia and their fluctuations through repeated clinical assessments using the Unified Dyskinesia Rating Scale - UDysRS
Dyskinesia | up to 1 month
  Evaluation of the performance of a wearable accelerometer in detecting dyskinesia (compared to patient reported dyskinesia in the patient diary)
"Time on" with and without dyskinesia | 1 month
  Evaluation of "time on" with and without dyskinesia, assessed through Patient Diary
"Time off" | 1 month
  Evaluation of "time off", assessed through Patient Diary
Patient controller usability | 1 month
  Usability will be evaluated by means of a usability questionnaire
Usability of the system for the physician | 1 month
  Usability will be evaluated by means of a usability questionnaire
Change in the TEED to the patient | 1 month
  Change in the Total Electrical Energy Delivered (TEED) to the patient

CONTACTS AND LOCATIONS:
Locations (8):
- Italy (5):
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - IRCCS Istituto Neurologico Carlo Besta, Milan
  - Azienda Ospedale Universitario di Padova - Università di Padova, Padua
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome
  - AOU Città della Salute e della Scienza di Torino, Turin
- Maastricht Medical Center, Maastricht, Netherlands
- Poland (2):
  - Copernicus Podmiot Leczniczy, Gdansk
  - Narodowy Instytut Onkologii im. Marii Skłodowskiej-Curie - Państwowy Instytut Badawczy, Warsaw

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Marceglia S, Conti C, Svanidze O, Foffani G, Lozano AM, Moro E, Volkmann J, Arlotti M, Rossi L, Priori A. Double-blind cross-over pilot trial protocol to evaluate the safety and preliminary efficacy of long-term adaptive deep brain stimulation in patients with Parkinson's disease. BMJ Open. 2022 Jan 3;12(1):e049955. doi: 10.1136/bmjopen-2021-049955. PMID 34980610